CLINICAL TRIAL: NCT05432856
Title: Impact of Metabolic Health Patterns And Breast Cancer Over Time in Women
Acronym: IMPACT-Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HREBA.CC-22-0128
Record Dates: First submitted 2022-06-10; First posted 2022-06-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Diseases; Cardiovascular Morbidity; Metabolic Disease
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Diseases | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-Restricted Eating and Sedentary Time Reduction (Experimental): Group 1 (Experimental intervention): Participants assigned to this group will receive standard chemotherapy treatment plus a dietary program, and sedentary time reduction strategies, program and a Fitbit monitor. If you are randomized into this group, you will be asked to follow TRE, will receive nutritional education and individualized recommendations on improving diet quality and healthy eating practices, and given to strategies to work towards reducing sedentary time. These components will be gradually introduced over the 24-week program.
  Interventions: Behavioral: Time restricted eating, nutrition education, and sedentary time reduction strategies
- Nutrition and Exercise Guidelines (No Intervention): Group 2 (Non-experimental intervention): Participants randomized to this group will receive standard chemotherapy treatment plus a single, group-based "nutrition during cancer" class, as well as a copy of Canada's Food Guide, physical activity guidelines, and a Fitbit monitor. You will be asked to only make dietary changes if they are recommended within the class or by your doctor, and to maintain your usual timing and number of meals consumed per day. Throughout the 24-week period, you will receive seven brief phone calls from a study staff member to ask about your symptoms and provide support. After the end of the study, participants in this group will be offered a one-one-one counselling session with a registered dietitian.

INTERVENTIONS:
Behavioral: Time restricted eating, nutrition education, and sedentary time reduction strategies — 1. TRE: You will be asked to eating as much as you like but only within an 8-10 hour window and then do not eat, or "fast" by consuming only water, black coffee or tea without milk/sugar for a window of 16 hours per day. This protocol will be required for 5 or more days in a row each week.
  2. Nutrition education and individualized recommendations: You will receive an assessment, and one-on-one education on healthy eating according to Canada's dietary guidelines, with individualized small goal each to improve your dietary habits.
  3. Sedentary time reduction: Using the provided Fitbit wrist monitor, you will be asked to track and gradually increase your daily step counts, break up periods of inactivity, and try to incorporate ways to decrease sedentary behaviour in everyday life.
  Arms: Time-Restricted Eating and Sedentary Time Reduction

SUMMARY:
Background & Rationale:

Breast cancer (BC) is the most commonly diagnosed malignancy in women worldwide (2.1 million diagnoses in 2018, 25% of new cancer cases). In Canada, early stage BC mortality rates have decreased by 48% over the past 30 years as a result of advances in prevention, detection, and treatment. However, competing risks for mortality from non-cancer causes have emerged, where cardiovascular disease (CVD) is now a leading cause of death for BC survivors. The direct toxic effects of BC treatment on the heart (cardiotoxicity) are well characterized by the investigators and many others, as a contributor to elevated cardiovascular risk. However, BC treatment and the associated lifestyle changes (i.e. physical inactivity, poor diet quality, stress) are increasingly recognized to also strongly affect metabolism negatively manifesting as insulin resistance, dyslipidemia and adipose tissue (fat) accumulation. These adverse metabolic changes are strongly linked to CVD risk and represent a currently underappreciated contributor to the elevated CVD risk among BC survivors. Preliminary data and recent publications demonstrate that regional fat accumulation occurs during BC treatment and that the fat burden in key locations is associated with poor cardiorespiratory health. A trigger of these adverse metabolic and inflammatory effects is excess fat specifically within ectopic fat (viscera, intermuscular, or hepatic) regions. In 2019, a member of the study team found that the volume of visceral and intermuscular but not subcutaneous fat at BC diagnosis were linearly associated with CVD events within 6 years, even among those with normal BMI and after adjustment for pre-existing CVD risk factors and for BC treatment type. Using MRI, investigators found that ~1 year after chemotherapy, BC survivors had significantly larger depots of visceral fat (49% larger) and thigh intermuscular fat (41% larger) compared to age and sex-matched controls, despite similar BMI and subcutaneous fat volumes in the two groups. Investigators also showed that the fat fraction within the thigh muscle and visceral fat volumes independently explained ~50% of the variation in cardiorespiratory fitness (measured by peak VO2). In particular, peak VO2 is one of the most powerful predictors of all-cause and CVD mortality and health care costs, and is the most consistently reported negative sequelae after treatment for BC. Unfortunately, there are no known therapies to recover long-term myocardial damage (i.e. cell death, fibrosis) from cancer therapies. There are several reasons to target fat as a therapeutic target in BC patients: 1) The study team have compelling preliminary data showing accelerated formation of ectopic fat during BC treatment. 2) Investigator's recent data showed that high fat content in key fat pools was associated with reduced peak VO2. 3) The burden of fat and the associated metabolic abnormalities are dynamic and malleable, and thus highly treatable.

Research Question & Objectives:

The primary purpose of this study is to evaluate the effect of a behavioural intervention involving supported time-restricted eating (TRE), diet quality improvements, and reduced sedentary time versus usual cancer and nutrition care in BC patients receiving chemotherapy treatment on ectopic fat, cardiometabolic profile, and chemotherapy outcomes. The investigators hypothesize that the intervention will attenuate the growth of ectopic fat during chemotherapy and reduce chemotherapy symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Female biological sex at birth
* >18 years
* Diagnosis of stage I, II, or III breast cancer
* starting neoadjuvant or adjuvant intravenous chemotherapy
* ECOG <3;
* Oncologist approval to participate;
* English speaking (all study materials and study staff will be in English)
* Willing and able to adhere to study intervention

Exclusion Criteria:

* Individuals who do not have access to a smart phone with Bluetooth capability (required for Fitbit and for responding to intervention text messages) or at least a shared cell phone with someone in the same household (i.e., some couples may share a phone).
* Type 1 or type 2 diabetes who require exogenous insulin (due to the potential need to adjust insulin dosing with TRE) or with hemoglobin A1c >10%
* Research MRI contraindications (e.g., pacemaker, magnetic implants, pregnancy)
* Uncontrolled thyroid disorder
* Self-reported eating disorder history
* Body mass index <18.5 kg/m2 or clinical signs of cachexia (discretion of treating oncologist)
* ≥5% body weight loss within last 6 months
* Those who are currently working night/rotating shifts, eating within ≤10-hour window or consistently eating less than 3 meals/day in the past 3 months.
* patients who meet the criteria for medical clearance prior to exercise using the Physical Activity Readiness Questionnaire+ and are not cleared by their treating oncologist or family physician to perform maximal exercise testing.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female biological sex at birth.
Enrollment: 65 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in Fat Volumes | Baseline, 24-weeks, and 2 years
  Visceral fat volumes as measured by MRI.

SECONDARY OUTCOMES:
Change in Thigh Fat Pool Volume | Baseline, 24-weeks, and 2 years
  Thigh intermuscular and intramuscular fat volumes as measured by MRI.
Change in Liver Fat Volume | Baseline, 24-weeks, and 2 years
  Volume of fat in the hepatocytes in the liver as measured by MRI.
Change in Subcutaneous Abdominal Fat Volume | Baseline, 24-weeks, and 2 years
  Subcutaneous fat volumes that surround the abdomen as measured by MRI.
Change in Metabolic Syndrome Z-score | Baseline, 24-weeks, and 2 years
  Defined by the National Cholesterol Education Program Adult Treatment Panel, metabolic syndrome is determined by the presence of 3 or more of the following: abdominal obesity defined by waist circumference (men >102cm, women >88cm), triglycerides ≥150mg/dL, fasting glucose ≥110mg/dL, HDL cholesterol <40mg/dL for men and <50mg/dL for women, and blood pressure of ≥130/≥85mmHg. Z-scores of 0 are equal to the mean. Anything above 0 for each risk listed above (excluding HDL cholesterol) indicates higher risk of CVD. Since HDL cholesterol is healthy, higher z-scores indicate lower risk of CVD. Z-scores rarely fall outside a range of -3 to 3.
Change in Framingham risk score | Baseline, 24-weeks, and 2 years
  Using the Framingham risk score to determine cardiovascular disease risk calculated using the Canadian Cardiovascular Society scoring system for age, sex, total cholesterol (mg/dL), high-density lipoprotein (mg/dL), treated or untreated systolic blood pressure (mmHg), diabetes, and smoking status (self-reported in questionnaires). Each category listed above is also assigned a numeric value. To find risk, one must total their points together from each category. The minimum value ranges from -3 or less points to a maximum value range of 21+ points. -3 or less points indicates a very low risk of cardiovascular disease, and 21+ points indicates a high risk of cardiovascular disease.
Change in Peak VO2 | Baseline, 24-weeks, and 2 years
  Maximal amount of oxygen consumed during a cardiopulmonary exercise test on a cycle ergometer measured by mL/kg/min to indicate cardiorespiratory fitness.

OTHER OUTCOMES:
Change in Insulin Resistance | Baseline, 24-weeks, and 2 years
  Using blood work to determine insulin resistance, this includes HOMA-IR (mg/dL), hemoglobin A1c (mg/dL), lipid profile (mg/dL), and fasting glucose (mg/dL).
Change in Waist to Hip ratio | Baseline, 24-weeks, and 2 years
  Measurement of abdominal circumference at the level of the umbilicus, recorded to the nearest 0.5 cm, and measurement of circumference of the hips to the nearest 0.5 cm to calculate waist-to-hip ratio.
Change in Resting Blood Pressure | Baseline, 24-weeks, and 2 years
  Manually measured using a stethoscope and sphygmomanometer in a seated position after five minutes of quiet rest. The average of 2 measurements, taken 60 seconds apart that are within 6 mmHg will be taken.
Change in Hormonal Markers | Baseline, 24-weeks, and 2 years
  Measure of leptin and adiponectin (hormones involved in fat regulation) in blood recorded in ng/mL and ug/mL respectively.
Medical Outcomes | Up to 10 years after study completion
  Descriptive data and chemotherapy outcomes, as well as tracking long-term health effects of participation through participants' electronic medical records.
Change in Cytokines | Baseline, 24-weeks, and 2 years
  Measure of cytokines IL-6 and TNF-a in blood recorded in pg/mL.
Physical Activity | through study completion, an average of 2 years
  Volume of time spent physically active measured by Fitbit Inspire 2 wrist band.
Dietary Intake | Up to 24 weeks
  Dietary intake will be assessed by 3-day food diary that is to be recorded over 2 consecutive weekdays and 1 weekend day, and will be collected using the Canadian version of the Automated Self-Administered 24-hour Dietary Assessment Tool (ASA24-Canada).
Smoking Status | Baseline
  Status as self-reported by participants in a qualitative demographics questionnaire. Participants may respond yes or no. Participants who smoke may indicate a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Thompson, PhD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - University of Toronto, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Information collected during the study will be used in analyses and will be published/ presented to the scientific community at meetings and in journals. In addition, study data without any identifying information will be shared with the research team at the University of Toronto, where the study is also taking place.